CLINICAL TRIAL: NCT02183337
Title: Relative Bioavailability of Both BI 1356 and Pioglitazone After Co-administration Compared to the Bioavailability of Multiple Oral Doses of BI 1356 10 mg qd Alone and Pioglitazone 45 mg qd Alone in Healthy Male and Female Volunteers (an Open Label, Randomised, Multiple-dose, Two-way Crossover Study)
Brief Title: Bioavailability of BI 1356 With and Without Co-administration of Pioglitazone and the Bioavailability of Pioglitazone With and Without Coadministration of BI 1356 in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.13
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Pioglitazone

ARMS (2):
- BI 1356 (Experimental): Treatment sequence AB_C or C_AB
  * Treatment A: 5 days BI 1356 until steady state followed by
  * Treatment B: combined treatment of BI 1356 with pioglitazone for 7 days
  * Treatment C: 7 days of treatment with Pioglitazone alone
  Interventions: Drug: BI 1356; Drug: BI 1356 + Pioglitazone; Drug: Pioglitazone
- Pioglitazone (Active Comparator): Treatment sequence AB_C or C_AB
  * Treatment A: 5 days BI 1356 until steady state followed by
  * Treatment B: combined treatment of BI 1356 with pioglitazone for 7 days
  * Treatment C: 7 days of treatment with Pioglitazone alone
  Interventions: Drug: BI 1356; Drug: BI 1356 + Pioglitazone; Drug: Pioglitazone

INTERVENTIONS:
Drug: BI 1356
Drug: BI 1356 + Pioglitazone
Drug: Pioglitazone

SUMMARY:
Study to investigate the bioavailability of BI 1356 with and without co-administration of pioglitazone and the bioavailability of pioglitazone with and without coadministration of BI 1356

ELIGIBILITY:
Inclusion Criteria:

* Healthy females and males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests
* Age ≥18 and Age ≤65 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections (e.g. HIV)
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsade de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

For male subjects:

* Not willing to use adequate contraception (condom use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, IUD [intrauterine device]) during the whole study period from the time of the first intake of study drug until one month after the last intake

For female subjects:

* Pregnancy or planning to become pregnant within 2 months of study completion
* Positive pregnancy test
* Are not willing or are unable to use a reliable method of contraception (such as implants, injectibles and combined oral contraceptives, sterilisation, IUD, double barrier method) for at least 3 months prior to participation in the trial, during and up to 2 months after completion/termination of the trial
* Chronic use of oral contraception or hormone replacement containing ethinyl estradiol as the only method of contraception
* Lactation period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 21 days
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 21 days

SECONDARY OUTCOMES:
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state) | up to 21 days
C24,ss (concentration of the analyte in plasma at steady state after administration of the last dose at the end of the dosing interval) | up to 21 days
λz,ss (terminal rate constant in plasma at steady state) | up to 21 days
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | up to 21 days
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | up to 21 days
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) | up to 21 days
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | up to 21 days
Changes in physical examination (including body weight) | up to 27 days after last administration of study medication
Changes in Vital signs (Blood pressure (BP), Pulse Rate (PR) | up to 27 days after last administration of study medication
Changes in 12-lead ECG (electrocardiogram) | up to 27 days after last administration of study medication
Changes in clinical laboratory values | up to 27 days after last administration of study medication
Number of patients with adverse events | up to 27 days after last administration of study medication
Assessment of tolerability by investigator on a 4-point scale | up to 27 days after last administration of study medication